CLINICAL TRIAL: NCT02482844
Title: Assessment of the Prognosis of Persistent Left Bundle Branch Block (LBBB) After Transcatheter Aortic Valve Implantation (TAVI ) by an Electrophysiological and Remote Monitoring Risk-adapted Algorithm
Brief Title: Assessment of the Prognosis of Persistent Left Bundle Branch Block (LBBB)After Transcatheter Aortic Valve Implantation (TAVI ) by an Electrophysiological and Remote Monitoring Risk-adapted Algorithm
Acronym: LBBB-TAVI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: LivaNova (Industry); Biotronik France (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: CHU-0239; 2015-A00271-48 (Registry Identifier: 2015-A00271-48)
Record Dates: First submitted 2015-06-18; First posted 2015-06-26 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Post-TAVI
Keywords: TAVI; de novo and persistent LBBB; electrophysiology; Holter; pacemaker

ARMS (2):
- Pacemaker (Other): Every patient included with a de novo LBBB, persistent that is observed beyond 24 hours after the TAVI procedure, will benefit from an endocavitary electrophysiological exploration . According to the meditative delay of conduction, we shall hold the setting-up of a pacemaker in case of delay lengthened HV (> 70 ms) or of infrahissian block, in the opposite case the implantation of an holter with remote monitoring will be made
  Interventions: Other: pacemaker implantation
- holter implantable (Other): Every patient included with a de novo LBBB, persistent that is observed beyond 24 hours after the TAVI procedure, will benefit from an endocavitary electrophysiological exploration . According to the meditative delay of conduction, we shall hold the setting-up of a pacemaker in case of delay lengthened HV (> 70 ms) or of infrahissian block, in the opposite case the implantation of an holter with remote monitoring will be made
  Interventions: Other: holter implantation

INTERVENTIONS:
Other: pacemaker implantation
  Arms: Pacemaker
Other: holter implantation
  Arms: holter implantable

SUMMARY:
The replacement of the aortic valve by percutaneous approach (called TAVI) is a therapy which is booming in the management of aortic stenosis. It concerns patients who have a high surgical risk presenting comorbidity, for whom a classic approach by surgery of valvular replacement seems unreasonable. Beyond its feasibility, the implantation of a TAVI is less invasive and improves the patient's morbi-mortality. The appearance of a Left Bundle Branch Block (LBBB) is one of the most frequent complications of this procedure and represents an important risk of atrio-ventricular (AV) high grade conductive disorders requiring permanent pacing in 5 in 15 % of the cases in 1 year.

De novo LBBB is associated with a more important morbi-mortality in post-TAVI situation. However, there are no predictive elements of these conductive disorders. Besides, the incidence and the deadline of appearance of this AV disorders are not established. It seems relevant to propose a new stratification based on ECG and endocavitary data. The monitoring of the conductive disorders is allowed by remote monitoring thanks to the implantation of a pacemaker or an implantable holter allowing to determine the incidence and the deadline of appearance of high grade AV conduction disorders.

DETAILED DESCRIPTION:
The aim of this protocol is to study the appearance of the high grade AV conductive disorders at 12 months by monitoring for patients with a de novo LBBB after TAVI from an adapated algorithm to the risk and based on an early electrophysiological evaluation.

The recruitment of patients takes place in each cardiology department. The project is submitted to the Ethics Committee .

The patients are informed about this study by the investigator. After a reflection period and an answer to the possible questions, the patient is included. The informed consent is signed.

Every patient included with a de novo LBBB, persistent that is observed beyond 24 hours after the TAVI procedure, will benefit from an endocavitary electrophysiological exploration . According to the meditative delay of conduction, a pacemaker will be implanted in case of delay lengthened HV (> 70 ms) or of infrahissian block, in the opposite case the implantation of an holter with remote monitoring will be made.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 year's old
* Patient implanted by a percutaneous biological aortic valve according to the recommendations of the European society of cardiology according to the guidelines of ESC 2012
* Life expectancy upper 1-year-old
* Sinusal rhythm
* Patient with a de novo LBBB post-TAVI persitent and observed beyond 24 hours after the procedure of TAVI.

Exclusion Criteria:

* Patient with a pacemaker pre-TAVI
* Patient with LBBB pre-procedure
* Pregnancy
* Permanent atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
To assess the aAppearance (rate and deadlinetime after TAVI) of AV high-grade conductive disorders (complete AV block and AV block II Mobitz 2) in patients with de novo LBBB induced by TAVI. | at 12 months

SECONDARY OUTCOMES:
To assess the appearance (rate and time after TAVI) of AV high-grade conductive disorders (complete AV block and AV block II Mobitz 2) in patients with de novo LBBB induced by TAVI | at 3 months and at 6 months
To identify predictive factors of AV high-grade conductive disorders in patients with de novo LBBB induced by TAVI | at 3 months, 6 months and 12 months
To assess impact of de novo LBBB induced by TAVI on mortality (cardiovascular, heart failure, all causes) and hospitalizations (cardiovascular, heart failure, all causes) | at 3 months, 6 months and 12 months
To assess safety (adverse events) of proposed management (endocardial electrophysiological study, permanent pacemaker implantation) in such patients | at 3 months, 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Romain ESCHALIER, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Massoullie G, Bordachar P, Irles D, Caussin C, Da Costa A, Defaye P, Jean F, Mechulan A, Mondoly P, Souteyrand G, Pereira B, Ploux S, Eschalier R. Prognosis assessment of persistent left bundle branch block after TAVI by an electrophysiological and remote monitoring risk-adapted algorithm: rationale and design of the multicentre LBBB-TAVI Study. BMJ Open. 2016 Oct 26;6(10):e010485. doi: 10.1136/bmjopen-2015-010485. PMID 27797979